CLINICAL TRIAL: NCT03902587
Title: Application of Cervical Elastography in Obstetrics
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 18-01598
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Cervical Elastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cervical Elastography: During each sonogram in which cervical lengths are measured, 5 additional cervical indices will be collected using Samsung's E-cervix technology. Each index will then be separated based on characteristics to create a nomogram for singletons, twins, and those with interventions already in place (i.e. cerclage and/or progesterone) at the time of their E-cervix assessment.
  Interventions: Device: Samsung's E-cervix technology

INTERVENTIONS:
Device: Samsung's E-cervix technology — While patients are having their routine cervical ultrasound assessments which requires a 5 minute time period, we will use the built-in software to obtain additional E-cervix measurements to evaluate the consistency of the cervical os. This will be done within the standard 5 minute period which is typically done to observe for dynamic changes. The measurements will be obtained with the same sonogram machine, using updated software.

SUMMARY:
The purpose of this study is to develop cervical elastography nomograms using Samsung's novel technology "E-cervix" and determine its ability to predict preterm birth.

During each sonogram in which cervical lengths are measured, 5 additional cervical indices will be collected using Samsung's E-cervix technology. Each index will then be separated based on characteristics to create a nomogram for singletons, twins, and those with interventions already in place (i.e. cerclage and/or progesterone) at the time of their E-cervix assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women who present for early screening or level II ultrasound, aged 18 to 50 years, provides written Informed consent and is willing to comply with protocol requirements, and obtained cervical length and measurements using the E-cervix software/hardware

Exclusion Criteria:

* >50 years old
* prior cervical surgical procedures (i.e. LEEP procedure, cold knife cone biopsy)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who present for early screening or level II ultrasound
Study Population: Women who present for early screening or level II ultrasound, aged 18 to 50 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Number of preterm Births | 24 Months

SECONDARY OUTCOMES:
E-cervix indices | 18 Weeks, 19 Weeks, 20 Weeks, 21 Weeks, 22 Weeks
  Pearson or Spearman correlation coefficients will be calculated to determine the association between the cervical length and each of the e-cervix parameters at the baseline assessment at 18-22 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Chavez, MD, Principal Investigator — NYU Winthrop Hospital
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Available upon request.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.